CLINICAL TRIAL: NCT03846401
Title: Evaluation of Role of Fiberoptic Bronchoscopy in Patients With Lower Respiratory Tract Infection in Respiratory Intensive Care Unit of Assiut University Hospital
Brief Title: Bronchoscopy in Lower Respiratory Tract Infection in Respiratory Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yara Yasser Omar, Chest Specialist in Assiut University Hospital, Assiut University
Other Study IDs: Bronchoscopy in LRTI
Record Dates: First submitted 2019-02-08; First posted 2019-02-19 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Lower Respiratory Tract Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: fiberoptic bronchoscopy — Will be performed according to British Thoracic Society guidelines 2013.
  -Microbiological methods The specimen (tracheal aspirate & BAL) will be collected under aseptic conditions in a sterile container and immediately sent to the laboratory for microbiological analyses.
  Samples will be apply for:
  1. Direct smear by Gram stain and ZeihlNelseen stain
  2. Samples culturedinBact/alert bottle(BioMérieux, France).
  3. Isolation of causative organism from positive cases by:
     Subculture on MacConkey , blood , chocolate agar , Sabouroud's agar and Lowenstien Jensen media.
  4. Identification of isolated organism and drug sensitivity test by Automated Vitek2 Compact(BioMérieux, France).
  5. Multiplex PCR for detection of Respiratory viruses in lower respiratory tract

SUMMARY:
Evaluate the diagnostic and therapeutic role of fiberoptic bronchoscopy in management of patients with lower respiratory tract infection in Respiratory Intensive Care Unit of Assiut University Hospital

DETAILED DESCRIPTION:
Since its introduction in daily medical practice in the late 20th century, fiberoptic bronchoscopy (FOB) has had an increasing role in the everyday life of the pulmonologist. Not only for diagnosis, but also for therapeutic interventions, it has achieved widespread use and is now performed in a diversity of clinical scenarios. For several reasons, from easy performance in trained hands to versatility, diagnostic reliability, and safety, flexible bronchoscopy is now widely accepted and increasingly used in the management of critically ill patients.

A wide range of indications exists for FOB in the intensive care unit (ICU). Most correspond to basic bronchoscopy with exploration, lavage, brushing, and forceps sampling as the primary used techniques. It is recommended that intensive care units account for the facility to perform urgent and timely FOB for a range of therapeutic and diagnostic purposes. Critical care settings demand that respiratory system problems be resolved and clinical decisions be made in a timely manner.

Although one can generally group the indications for bronchoscopy into diagnostic and therapeutic, there are circumstances in which the examination serves both purposes. The main indications for flexible bronchoscopy in the intensive care unit are the visualization of the airways, sampling for diagnostic purposes and management of the artificial airways.

Respiratory infections account for significant morbidity, mortality, and healthcare-related expenditure in patients admitted to the Intensive Care Unit (ICU). Respiratory infections account for 3.5 million deaths worldwide and 79 million loss of disability-adjusted life-years.

The bacteriological profile of pulmonary infections varies within the same country, with time due to differences in the frequency of use of antibiotics, environmental factors, and ventilation in the critically ill patients. Likewise, an expanded variety of emerging pathogens provide challenges for the microbiology laboratory. It has been reported clinical microbiologists in diagnostic laboratories have a critical role to play in the diagnosis and management of lower respiratory tract infection (LRTI) as overtreatment of acute uncomplicated pulmonary infections led to unparalleled levels of multi drug resistance among pathogens. Since the etiological agents of pulmonary infections (LRTI) cannot be determined clinically, microbial investigation is required for both treatment and management of individual case and for epidemiological purposes. Bronchoalveolar lavage (BAL) is an ideal sample that allows the recovery of pathogens cellular and non-cellular components from the epithelial surface of lower respiratory tract. Bronchoalveolar lavage has improved sensitivity and specificity of diagnostic techniques in diagnosis of pulmonary infection. It is increasingly utilized as diagnostic tool though in the past it remained as investigative and research tool as the sputum culture yields diagnosis in fewer than 50% of patients with pulmonary infections. Early diagnosis and proper choice of antimicrobials is crucial for management of these patients. The advent of bronchoscopy and quantitative analysis of BAL have improved sensitivity and specificity in diagnosis of pulmonary infections.

Antibiotics form the main stay of treatment of various respiratory infections which are often initiated empirically based on their previous experiences, hence, leading to the inappropriate use of antibiotics and antimicrobial resistance. Resistance to antibiotics has emerged recently due to misuse of antibiotics and is a threat to health-care system, especially in developing countries where there are no antimicrobial stewardship programs in most ICUs.

Antimicrobial resistance results in increased economic burden on patients due to the higher cost of antibiotics, prolonged ICU stay, and increased mortality. Prescribing appropriate antibiotics for the right duration is very important to prevent drug resistance. Local knowledge regarding the most common organisms and their resistance pattern in various infections will greatly assist clinicians in choosing appropriate initial antibiotic therapy. Hence, it is important to know the antibiotic prescribing pattern and resistance patterns in ICU.

In critically ill patients, mechanical ventilation might cause ventilator-induced lung injury and hospital-acquired pneumonia, both conditions promote atelectasis and stagnant secretions that may worsen oxygenation and delay weaning from ventilator.

Atelectasis may result from numerous causes, for example, from congestion of mucus in the central airways, from increased sputum production, from decreased mucociliary clearance, from decreased cough effectiveness, from increased sputum viscosity, or by a combination of these factors. Treatment of atelectasis in intensive care unit (ICU) patients has been focused on blind airway suctioning, bronchoscopy with or without adjuncts such as nebulization of N-acetylcysteine, and chest physiotherapy. Bronchoscopy is regarded as an attractive method for endobronchial mucus clearing, which possibly results in a more effective airway clearance as it is performed under direct visualization of the airways.

Therefore, removing the sputum is important for patient management, but blind negative pressure aspiration can damage the airway mucosa and leave sputum in place, worsening the patient's condition. Removing sputum under bronchoscopy could allow the precise removal of all sputum while minimizing mucosa damage.

Acute respiratory failure (ARF) has long been a challenge for physicians who perform bronchoscopy for diagnostic or therapeutic purposes. Hypoxaemia is aggravated when implementing bronchoalveolar lavage (BAL) or therapeutic intervention. Many physicians lose their chance to perform bronchoscopy and acquire adequate samples for appropriate treatment. Since undergoing a bronchoscopy can be hazardous to patients with ARF, intubation is preferred and physicians are reluctant to achieve BAL sample. Therefore, bronchoscopic procedures in high-risk patients, especially those with hypoxaemia, have long been a challenge in this field. Few clinical studies have shown the effectiveness of performing bronchoscopy using high flow nasal cannula (HFNC) in ARF for diagnostic purpose.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years old in R.I.C.U who are on mechanical ventilator or high flow nasal cannula oxygen with lower respiratory tract infection or who show atelectasis on CXR in which the standard therapy failed will be included in this study

Exclusion Criteria:

* Severely hypoxemic patients under high-FiO2 support and/or high PEEP, if the patient is unable to keep oxygen saturation >90% with an FiO2 of 0.9-1.0 or a PaO2/FiO2 ratio of <100, Severe acidosis, Ph<7,2
* Presence of pneumothorax
* Active bronchospasm.
* Patients with acute coronary problems, such as acute arrhythmia, acute myocardial infarction or ongoing hemodynamic instability, under vasoactive therapy.
* patients with known intracranial hypertension
* patients have coagulation abnormalities, such as thrombocytopenia or elevated prothrombin time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with lower respiratory tract infection in the Respiratory Intensive Care Unit (R.I.C.U.), Department of Chest Diseases and Tuberculosis, Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Antimicrobial resistance pattern | 1 year
  isolated organism and drug sensitivity test by Automated Vitek2 Compact(BioMérieux, France).

SECONDARY OUTCOMES:
pathogen identification | 1 year
  by Multiplex PCR
recovering an array of microorganisms | 1 year
  by BACT/ALERT® Culture Media

CONTACTS AND LOCATIONS:
Overall Officials: Maha K. Ghanem, Prof, Study Chair — Assiut University; Hoda A. Makhlouf, Prof, Study Director — Assiut University; Ali A. Hasan, ass. prof., Study Director — Assiut University; Asmaa O. Ahmed, ass. prof, Study Director — Assiut University

REFERENCES:
- [Background] Mahendra M, Jayaraj BS, Lokesh KS, Chaya SK, Veerapaneni VV, Limaye S, Dhar R, Swarnakar R, Ambalkar S, Mahesh PA. Antibiotic Prescription, Organisms and its Resistance Pattern in Patients Admitted to Respiratory ICU with Respiratory Infection in Mysuru. Indian J Crit Care Med. 2018 Apr;22(4):223-230. doi: 10.4103/ijccm.IJCCM_409_17. PMID 29743760
- [Background] Ahmed SM, Jakribettu RP, Meletath SK, B A, Vpa S. Lower Respiratory Tract Infections (LTRIs): An Insight into the Prevalence and the Antibiogram of the Gram Negative, Respiratory, Bacterial Agents. J Clin Diagn Res. 2013 Feb;7(2):253-6. doi: 10.7860/JCDR/2013/5308.2740. Epub 2013 Jan 10. PMID 23543819
- [Background] Jaffal K, Six S, Zerimech F, Nseir S. Relationship between hyperoxemia and ventilator associated pneumonia. Ann Transl Med. 2017 Nov;5(22):453. doi: 10.21037/atm.2017.10.15. PMID 29264370
- [Background] Smeijsters KMG, Bijkerk RM, Daniels JMA, van de Ven PM, Girbes ARJ, Heunks LMA, Spijkstra JJ, Tuinman PR. Effect of Bronchoscopy on Gas Exchange and Respiratory Mechanics in Critically Ill Patients With Atelectasis: An Observational Cohort Study. Front Med (Lausanne). 2018 Nov 13;5:301. doi: 10.3389/fmed.2018.00301. eCollection 2018. PMID 30483505
- [Background] Qiao Z, Yu J, Yu K, Zhang M. The benefit of daily sputum suction via bronchoscopy in patients of chronic obstructive pulmonary disease with ventilators: A randomized controlled trial. Medicine (Baltimore). 2018 Aug;97(31):e11631. doi: 10.1097/MD.0000000000011631. PMID 30075543
- [Background] Chung SM, Choi JW, Lee YS, Choi JH, Oh JY, Min KH, Hur GY, Lee SY, Shim JJ, Kang KH. Clinical Effectiveness of High-Flow Nasal Cannula in Hypoxaemic Patients during Bronchoscopic Procedures. Tuberc Respir Dis (Seoul). 2019 Jan;82(1):81-85. doi: 10.4046/trd.2017.0104. Epub 2018 Jun 19. PMID 29926544